CLINICAL TRIAL: NCT00771927
Title: Post-Authorization Safety Study to Evaluate the Long-Term Safety and Tolerability of Vimpat® (Lacosamide) as Add-On Therapy in Epilepsy Patients With Partial-Onset Seizures Who Are Uncontrolled on Current Therapy
Brief Title: Post-Authorization Safety Study to Assess the Safety of Vimpat as add-on Therapy in Patients With Partial-onset Seizures
Acronym: PASS
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SP0942
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2013-05

CONDITIONS: Epilepsies, Partial
Keywords: Vimpat®; Lacosamide; LCM; epilepsy; epilepsies; seizure; partial seizure; partial onset; seizure disorder; single seizure; motor seizure; convulsions; add-on; AED; anti-epileptic; anti-epileptic drug; seizure control; open-label; post authorization; PASS; late stage; trial; study; phase 4; phase IV
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lacosamide: Epilepsy patients with partial-onset seizures who are uncontrolled on current therapy and are treated with add-on Vimpat
  Interventions: Drug: Lacosamide
- Other AED: Epilepsy patients with partial-onset seizures who are uncontrolled on current therapy and are treated with other approved AED as add-on therapy

INTERVENTIONS:
Drug: Lacosamide — Vimpat was used as per site routine practices, and in-line with the marketing authorization.
  Other Names: Vimpat®
  Groups: Lacosamide

SUMMARY:
SP942 is a non-interventional post-authorization safety study (PASS) to evaluate the long-term safety and tolerability of Vimpat® (Lacosamide, LCM) as add-on treatment in patients with Epilepsy 16 years and older with partial-onset seizures who are uncontrolled on current therapy. Using reported adverse events, the incidence of certain cardiovascular and psychiatric events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* This study includes any subject 16 years or older who has an Epilepsy diagnosis with Partial-Onset Seizures; and whose Seizure activity is uncontrolled on current therapy
* Patients who are prescribed Vimpat or any other add-on Antiepileptic Drug (AED) may be included in the study
* The initiation of an add-on AED therapy can not be more than 2 days before the patient's start of the study

Exclusion Criteria:

* N/A

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Institutions, hospitals, primary care clinics and community based
Sampling Method: Non-Probability Sample
Enrollment: 1005 (Actual)
Dates: Start 2008-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (62):
- France (8):
  - Bron
  - Dijon
  - La Tronche
  - Montpellier
  - Nantes
  - Paris
  - Saint-Brieuc
  - Tain-l'Hermitage
- Germany (35):
  - Aschaffenburg
  - Bad Berka
  - Berlin
  - Bernau
  - Bielefeld
  - Bonn
  - Dresden
  - Düsseldorf
  - Erlangen
  - Essen
  - Freiburg im Breisgau
  - Göttingen
  - Halle
  - Hamburg
  - Jena
  - Kehl-Kork
  - Kiel
  - Koningstein-Falkenstein
  - Krefeld
  - Mainz
  - Marburg
  - München
  - Münster
  - Neuburg am Inn
  - Neukirchen-Vluyn
  - Oldenburg
  - Osnabrück
  - Potsdam
  - Radeberg, Sachsen
  - Ravensburg
  - Rotenburg (Wümme)
  - Stuttgart
  - Ulm
  - Vogtareuth
  - Westerstede
- Netherlands (3):
  - Blaricum
  - Heeze
  - Nijmegen
- Spain (2):
  - Barcelona
  - El Vendrell
- United Kingdom (14):
  - Plymouth, Devon
  - Fulwood, Preston, Lancashire
  - Bangor
  - Birmingham
  - Cardiff
  - Dundee
  - Edinburgh
  - Leeds
  - Leicester
  - London
  - Middlesbrough
  - Salford
  - Sheffield
  - Stoke-on-Trent

REFERENCES:
- See also: Product information — http://www.vimpat.com/pdf/PI.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled into 1 of 2 groups in this study (500 unique patients per group) at the discretion of the treating physician: patients treated with Vimpat as add-on to their current Anti-Epileptic Drug (AED) therapy (group 1) and patients treated with other approved AEDs as add-on (group 2).
Pre-assignment Details: Patient procedures and assessments were performed in the frame of the current standard practice at the discretion of the treating physician. Each patient was followed for the initial 12 months of add-on AED treatment. A Safety Follow-Up Visit is recommended for any patient who terminates add-on AED treatment before the end of the study period.
Period: Overall Study
Arm/Group | Lacosamide | Other AED
Started | 511 (Participant Flow and Baseline Characteristics refer to the Safety Set population.) | 493 (Participant Flow and Baseline Characteristics refer to the Safety Set population.)
Completed | 256 | 256
Not Completed | 255 | 237
Not completed — Adverse Event | 100 | 105
Not completed — Lack of Efficacy | 70 | 42
Not completed — Lost to Follow-up | 46 | 46
Not completed — Withdrawal by Subject | 16 | 17
Not completed — Other reason | 23 | 27

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Safety Set (SS). Safety Set includes all patients who have signed a data consent form, provided Baseline characteristic data, and received treatment at least once.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide | Other AED | Total
Number analyzed (Participants) | 511 | 493 | 1004
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 14 | 34
  Between 18 and 65 years | 467 | 434 | 901
  >=65 years | 24 | 45 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (13.58) | 42.3 (15.38) | 41.0 (14.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 282 | 548
  Male | 245 | 211 | 456
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 481 | 464 | 945
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 24 | 22 | 46
Weight [Mean (Standard Deviation); unit: kilogram] | 75.5 (18.10) | 75.7 (17.68) | 75.6 (17.89)
Height [Mean (Standard Deviation); unit: centimeter] | 170.4 (10.97) | 169.5 (9.24) | 170.0 (10.18)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 26.0 (5.89) | 26.2 (5.25) | 26.1 (5.59)

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Predefined Cardiovascular Treatment-Emergent Adverse Events (TEAEs) in Epilepsy Patients With Partial-onset Seizures While on Vimpat or Any Other add-on Antiepileptic Drug (AED) Treatment During the Study
Description: Predefined cardiovascular-related Adverse Events (AEs), ie, Atrioventricular (AV) block, syncope, bradycardia, and PR prolongation, were identified as AEs coded to one of the following MedDRA Preferred Terms: Adams-Stokes syndrome, Atrioventricular block, Atrioventricular block complete, Atrioventricular block first degree, Atrioventricular block second degree, Syncope, Bradycardia, Bradyarrhythmia, Sinus bradycardia, or Electrocardiogram PR prolongation.
  Treatment-emergent Adverse Events (TEAEs) are those that start on or after the day of first intake of the add-on AED treatment and up to 30 days after the day of last add-on AED treatment intake.
Time Frame: From Baseline up to 12 months
Population: Safety Set (SS) population
Measure: Number; unit: Treatment-Emergent Adverse Events
Arm/Group | Lacosamide | Other AED
Number analyzed (Participants) | 511 | 493
Treatment-Emergent Adverse Events | 4 | 3

2. Secondary Outcome: The Incidence of Predefined Psychiatric Treatment-Emergent Adverse Events (TEAEs) in Epilepsy Patients With Partial-onset Seizures While on Vimpat or Any Other add-on Antiepileptic Drug (AED) Treatment During the Study
Description: Predefined psychiatric-related AEs, ie, depression, suicide/self-injury, drug abuse, drug dependence, substance abuse, and intentional drug misuse were predefined as AEs coded to one of the following MedDRA Preferred Terms: Depression, Major depression, Depressed mood, Depression suicidal, Completed suicide, Suicidal behavior, Suicidal ideation, Suicide attempt, Intentional self-injury, Self-injurious behavior, Self-injurious ideation, Poisoning deliberate, Drug abuse, Drug abuser, Drug dependence, Substance abuse, Substance abuser, Polysubstance dependence, Intentional drug misuse, Intentional overdose, or Multiple drug overdose intentional.
  Treatment-emergent Adverse Events (TEAEs) are those that start on or after the day of first intake of the add-on AED treatment and up to 30 days after the day of last add-on AED treatment intake.
Time Frame: From Baseline up to 12 months
Population: Safety Set (SS) population
Measure: Number; unit: Treatment-Emergent Adverse Events
Arm/Group | Lacosamide | Other AED
Number analyzed (Participants) | 511 | 493
Treatment-Emergent Adverse Events | 22 | 31

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the whole study from Baseline (Month 0) up to Visit 5 (Month 12).
Description: Adverse Events refer to the Safety Set (SS). SS includes all patients who have signed a data consent form, provided Baseline characteristic data, and received treatment at least once.
Arm/Group | Lacosamide | Other AED
Serious Adverse Events (participants affected / at risk) | 78/511 | 64/493
Other Adverse Events (participants affected / at risk) | 359/511 | 299/493
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=511) | Other AED (N=493)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Atrial Flutter (Cardiac disorders) | 2 (2) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (2)
Left Ventricular Failure (Cardiac disorders) | 0 (0) | 1 (1)
Foetal Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal Disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cyst Rupture (General disorders) | 1 (1) | 0 (0)
Drug Ineffective (General disorders) | 1 (1) | 0 (0)
Gait Disturbance (General disorders) | 1 (1) | 0 (0)
Idiosyncratic Drug Reaction (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden Unexplained Death in Epilepsy (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Brain Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular Graft Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-Traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Electroencephalogram (Investigations) | 1 (1) | 0 (0)
Weight Increased (Investigations) | 1 (1) | 0 (0)
Investigation (Investigations) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Malignant Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 16 (18) | 17 (21)
Epilepsy (Nervous system disorders) | 7 (7) | 3 (3)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1)
Grand Mal Convulsion (Nervous system disorders) | 3 (3) | 11 (12)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Status Epilepticus (Nervous system disorders) | 3 (3) | 1 (1)
Seizure Cluster (Nervous system disorders) | 2 (4) | 1 (1)
Ataxia (Nervous system disorders) | 1 (2) | 0 (0)
Balance Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Complex Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Partial Seizures (Nervous system disorders) | 1 (1) | 5 (8)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Temporal Lobe Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Toxic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1)
Postictal Paralysis (Nervous system disorders) | 0 (0) | 1 (2)
Psychomotor Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Emotional Disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 2 (2) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Conversion Disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Disturbance in Social Behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Generalised Anxiety Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Somatoform Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Expressive Language Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Personality Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion Induced (Surgical and medical procedures) | 1 (1) | 0 (0)
Brain Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Abscess Drainage (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=511) | Other AED (N=493)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 2 (2) | 0 (0)
Bundle Branch Block Right (Cardiac disorders) | 2 (2) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular Exrasystoles (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular Block First Degree (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Conduction Disorder (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Extrasystoles (Cardiac disorders) | 1 (1) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Bundle Branch Block Left (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 44 (49) | 11 (12)
Eustachian Tube Disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vestibular Disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
External Ear Inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 52 (61) | 18 (19)
Vision Blurred (Eye disorders) | 18 (18) | 13 (13)
Visual Impairment (Eye disorders) | 9 (9) | 2 (2)
Accomodation Disorder (Eye disorders) | 1 (1) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Excessive Eye Blinking (Eye disorders) | 1 (1) | 0 (0)
Eye Disorder (Eye disorders) | 1 (1) | 0 (0)
Eye Haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Eye Pain (Eye disorders) | 1 (1) | 1 (1)
Eye Swelling (Eye disorders) | 1 (1) | 0 (0)
Ocular Discomfort (Eye disorders) | 1 (1) | 0 (0)
Oscillopsia (Eye disorders) | 1 (1) | 0 (0)
Saccadic Eye Movement (Eye disorders) | 1 (1) | 0 (0)
Abnormal Sensation in Eye (Eye disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Exophthalmos (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (1)
Retinal Infarction (Eye disorders) | 0 (0) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 47 (49) | 23 (24)
Vomiting (Gastrointestinal disorders) | 15 (16) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 15 (15)
Constipation (Gastrointestinal disorders) | 6 (6) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 4 (4) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (5) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Flatulence (Gastrointestinal disorders) | 2 (2) | 3 (4)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Aphthous Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue Spasm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coeliac Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival Hyperplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 81 (93) | 61 (65)
Irritability (General disorders) | 11 (12) | 13 (14)
Gait Disturbance (General disorders) | 8 (9) | 8 (8)
Asthenia (General disorders) | 4 (5) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 0 (0)
Oedema Peripheral (General disorders) | 2 (2) | 4 (4)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1)
Implant Site Pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Spinal Pain (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Drug Therapeutic Incompability (General disorders) | 0 (0) | 1 (1)
Feeling Abnormal (General disorders) | 0 (0) | 2 (2)
Feeling Cold (General disorders) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Temperature Intolerance (General disorders) | 0 (0) | 1 (1)
Hepatic Pain (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (8) | 11 (13)
Influenza (Infections and infestations) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (4) | 0 (0)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
H1N1 Influenza (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter Gastritis (Infections and infestations) | 1 (1) | 0 (0)
Infected Bites (Infections and infestations) | 1 (1) | 0 (0)
Intraspinal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2)
Vaginal Infection (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Rash Pustular (Infections and infestations) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Tooth Abscess (Infections and infestations) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 3 (3)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 8 (8) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 3 (4)
Laceration (Injury, poisoning and procedural complications) | 4 (5) | 2 (2)
Ligament Sprain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Burns Third Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nail Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Open Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight Increased (Investigations) | 16 (16) | 8 (9)
Weight Decreased (Investigations) | 5 (5) | 12 (12)
Electrocardiogram QT Prolonged (Investigations) | 3 (3) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 1 (1)
Electroencephalogram (Investigations) | 2 (2) | 0 (0)
Blood Cholesterol Increased (Investigations) | 1 (1) | 0 (0)
Blood Glucose Abnormal (Investigations) | 1 (1) | 0 (0)
Blood Pressure Decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram Q Wave Abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST Segment Elevation (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T Wave Inversion (Investigations) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 2 (2)
Neurological Examination (Investigations) | 1 (1) | 0 (0)
Neurological Examination Abnormal (Investigations) | 1 (1) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 (0) | 1 (1)
Blood Calcium Decreased (Investigations) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1)
C-Reactive Protein Increased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram Low Voltage (Investigations) | 0 (0) | 1 (1)
Investigation (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (4) | 10 (11)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactose Intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Iron Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Posture Abnormal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis Stenosans (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Anorectal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 108 (129) | 45 (49)
Headache (Nervous system disorders) | 53 (57) | 26 (30)
Convulsion (Nervous system disorders) | 21 (21) | 15 (18)
Tremor (Nervous system disorders) | 20 (24) | 12 (15)
Ataxia (Nervous system disorders) | 16 (17) | 8 (8)
Memory Impairment (Nervous system disorders) | 16 (16) | 14 (14)
Somnolence (Nervous system disorders) | 14 (16) | 7 (7)
Aphasia (Nervous system disorders) | 11 (11) | 12 (12)
Balance Disorder (Nervous system disorders) | 10 (11) | 4 (4)
Disturbance in Attention (Nervous system disorders) | 8 (8) | 8 (8)
Nystagmus (Nervous system disorders) | 6 (9) | 0 (0)
Paraesthesia (Nervous system disorders) | 6 (6) | 12 (12)
Cognitive Disorder (Nervous system disorders) | 5 (5) | 5 (5)
Lethargy (Nervous system disorders) | 4 (4) | 1 (1)
Migraine (Nervous system disorders) | 4 (4) | 2 (2)
Speech Disorder (Nervous system disorders) | 4 (4) | 4 (4)
Amnesia (Nervous system disorders) | 3 (3) | 1 (1)
Epilepsy (Nervous system disorders) | 3 (4) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 0 (0)
Aura (Nervous system disorders) | 2 (2) | 0 (0)
Coordination Abnormal (Nervous system disorders) | 2 (2) | 0 (0)
Grand Mal Convulsion (Nervous system disorders) | 2 (2) | 3 (4)
Partial Seizures (Nervous system disorders) | 2 (5) | 1 (1)
Cerebellar Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Complex Partial Seizures (Nervous system disorders) | 1 (1) | 2 (3)
Cubital Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Dysgraphia (Nervous system disorders) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0)
Formication (Nervous system disorders) | 1 (1) | 0 (0)
Hypertonia (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Poor Quality Sleep (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor Hyperactivity (Nervous system disorders) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 1 (1)
Simple Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Altered State of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Depressed Level of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Drug Withdrawal Convulsions (Nervous system disorders) | 0 (0) | 1 (1)
Head Titubation (Nervous system disorders) | 0 (0) | 2 (2)
Hypokinesia (Nervous system disorders) | 0 (0) | 2 (2)
Intention Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Motor Dysfunction (Nervous system disorders) | 0 (0) | 1 (1)
Myoclonic Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve Compression (Nervous system disorders) | 0 (0) | 1 (1)
Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1)
Periodic Limb Movement Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Petit Mal Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Postictal Headache (Nervous system disorders) | 0 (0) | 1 (1)
Psychomotor Skills Impaired (Nervous system disorders) | 0 (0) | 2 (2)
Seizure Cluster (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Tension Headache (Nervous system disorders) | 0 (0) | 1 (1)
Vascular Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1)
Visual Field Defect (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 13 (13) | 20 (23)
Insomnia (Psychiatric disorders) | 13 (14) | 15 (15)
Aggression (Psychiatric disorders) | 8 (8) | 20 (20)
Anxiety (Psychiatric disorders) | 8 (9) | 6 (6)
Sleep Disorder (Psychiatric disorders) | 6 (6) | 11 (12)
Restlessness (Psychiatric disorders) | 5 (5) | 4 (4)
Depressed Mood (Psychiatric disorders) | 4 (4) | 5 (5)
Abnormal Behaviour (Psychiatric disorders) | 3 (3) | 0 (0)
Agitation (Psychiatric disorders) | 3 (3) | 3 (3)
Confusional State (Psychiatric disorders) | 3 (3) | 6 (6)
Mood Altered (Psychiatric disorders) | 3 (3) | 3 (3)
Affect Lability (Psychiatric disorders) | 2 (2) | 0 (0)
Bradyphrenia (Psychiatric disorders) | 2 (2) | 1 (1)
Mood Swings (Psychiatric disorders) | 2 (2) | 8 (9)
Nightmare (Psychiatric disorders) | 2 (2) | 1 (1)
Personality Disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 1 (2) | 0 (0)
Affective Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1) | 1 (1)
Drepressive Symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 1 (1)
Dyssomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysthymic Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 1 (1)
Impaired Reasoning (Psychiatric disorders) | 1 (1) | 0 (0)
Listless (Psychiatric disorders) | 1 (1) | 0 (0)
Loss of Libido (Psychiatric disorders) | 1 (1) | 0 (0)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Nocturnal Fear (Psychiatric disorders) | 1 (1) | 0 (0)
Reading Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Somatoform Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 1 (1)
TIC (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Decreased Activity (Psychiatric disorders) | 0 (0) | 1 (1)
Emotional Disorder (Psychiatric disorders) | 0 (0) | 4 (4)
Food Aversion (Psychiatric disorders) | 0 (0) | 2 (2)
Initial Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Libido Decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Panic Attack (Psychiatric disorders) | 0 (0) | 1 (1)
Panic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Postictal Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition Frequency Decreased (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Menstrual Disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Menopausal Disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (12) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 8 (8) | 10 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6)
Heat Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Amygdalohippocampectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Brain Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Drug Therapy Changed (Surgical and medical procedures) | 1 (1) | 0 (0)
Intervertebral Disc Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth Extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Uterine Dilation and Curettage (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Vagal Nerve Stimulator Implantation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)
Hot Flush (Vascular disorders) | 2 (2) | 1 (1)
Circulatory Collapse (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 4 (4)
Venous Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Coldness (Vascular disorders) | 0 (0) | 2 (2)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Folate Deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days